CLINICAL TRIAL: NCT00255983
Title: Prospective, Randomized, Double-Blind Trial to Evaluate the Efficacy and Safety of Faropenem Medoxomil 600 mg PO, BID for 5 Days Versus Placebo In the Treatment of Acute Exacerbation of Chronic Bronchitis
Brief Title: A Trial to Evaluate the Efficacy and Safety of Faropenem Medoxomil In the Treatment of Chronic Bronchitis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: financial reasons
Sponsor: Replidyne (Industry)
Collaborators: INC Research Limited (Industry)
Responsible Party: Robert Tosiello, Replidyne
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REP-FAR-005
Record Dates: First submitted 2005-11-16; First posted 2005-11-21 (Estimated); Last update posted 2008-06-03 (Estimated); Status verified 2008-05

CONDITIONS: Chronic Bronchitis
Keywords: bronchitis; AECB
MeSH Terms: conditions — Bronchitis, Chronic; Bronchitis | interventions — faropenem medoxomil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): faropenem medoxomil
  Interventions: Drug: Faropenem medoxomil
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Faropenem medoxomil — 600 mg BID for 5 days
  Arms: 1
Drug: placebo — placebo tablets BID for 5 days
  Arms: 2

SUMMARY:
Identifying the role of antibiotics in the treatment of subjects with a microbiologically documented acute exacerbation of chronic bronchitis (AECB) is the purpose of this clinical trial. The trial has been designed to evaluate the efficacy and safety of faropenem medoxomil versus placebo in the treatment of subjects with microbiologically documented AECB.

DETAILED DESCRIPTION:
This is a multi-center, multi-national, prospective, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety/tolerability of faropenem medoxomil versus placebo in the treatment of subjects with a primary diagnosis of AECB. All subjects will have a pre-therapy sputum specimen obtained for culture and susceptibility testing.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female outpatients age greater than or equal 35 years with significant COPD (GOLD criteria I, IIA or IIB), chronic cough and sputum production and an acute exacerbation

Exclusion Criteria:

* Gold criteria III

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 491 (Actual)
Dates: Start 2005-12; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
• Clinical response at test of cure. | Day 8 to 12

CONTACTS AND LOCATIONS:
Overall Officials: Roger M Echols, MD, Study Director — Replidyne, Inc.
Locations (1):
- Multicenter, New Hope, Pennsylvania, United States